CLINICAL TRIAL: NCT04824352
Title: Apatinib in Combination With Ifosfamide and Etoposide (IE) for Relapsed or Refractory Osteosarcoma Progressed Upon First-line Chemotherapy (AIEO): a Prospective, Multiple-centre, Single-arm, Phase 2 Trial
Brief Title: Apatinib Plus IE Chemotherapy (Ifosfamide and Etoposide) for Relapsed or Refractory Osteosarcoma
Acronym: AIEO
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Because we then tried another trial with radomised design.
Sponsor: Peking University People's Hospital (Other)
Collaborators: Peking University Shougang Hospital (Other)
Responsible Party: Principal Investigator, Xie Lu, Musculoskeletal Tumor Center, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PKUPH-sarcoma 10
Record Dates: First submitted 2021-03-27; First posted 2021-04-01 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Effect of Drug; Toxicity, Drug
Keywords: osteosarcoma; apatinib; ifosfamide; etoposide; advanced
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Osteosarcoma | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- apatinib+IE (Experimental): Apatinib: 500 mg QD po (BSA ≥ 1.0) or 250 mg QD po (BSA < 1.0); IE: ifosfamide 1.8 g/m2/d d1-3; etoposide 100 mg/m2/d d1-3 Q2w
  Interventions: Drug: apatinib

INTERVENTIONS:
Drug: apatinib — Apatinib: 500 mg QD po (BSA ≥ 1.0) or 250 mg QD po (BSA < 1.0); IE: ifosfamide 1.8 g/m2/d d1-3; etoposide 100 mg/m2/d d1-3 Q2w
  Other Names: IE chemotherapy

SUMMARY:
Apatinib has led to positive responses in the treatment of osteosarcoma refractory to first-line chemotherapy. However, apatinib demonstrates only short-lived activity, and the disease control of musculoskeletal lesions is worse than that of pulmonary lesions. This treatment failure has been partly overcome by the addition of ifosfamide and etoposide (IE). We have ever retrospectively compared the activity of apatinib + IE in relapsed or refractory osteosarcoma in two sarcoma centers in China and concluded that for osteosarcoma with multiple sites of metastasis, apatinib + IE demonstrated clinically meaningful antitumor activity and delayed disease progression in patients with recurrent or refractory osteosarcoma after failure of chemotherapy. However to overcome the influence of other interventions on the outcome, we are currently performing a prospective trial to investigate this combination, from which more accurate data on this treatment strategy are expected.

ELIGIBILITY:
Inclusion Criteria:

* 1) histologically confirmed high-grade osteosarcoma;
* 2) initial treatment in the Orthopedic/Oncology Departments of Peking University People's Hospital or Peking University Shougang Hospital;
* 3) progression less than 6 months after first-line chemotherapy with a combination of high-dose methotrexate, doxorubicin, cisplatin and ifosfamide (first-line chemotherapy);
* 4) measurable lesions according to the Response Evaluation Criteria for Solid Tumors (RECIST 1.1) ;
* 5) Eastern Cooperative Oncology Group performance status ≤ 2 ;
* 6) acceptable haematologic, hepatic, and renal function.

Exclusion Criteria:

* those who had been previously treated with antiangiogenic TKIs and single IE chemotherapy;
* those who had severe or uncontrolled medical disorders that could jeopardize the outcomes of the study. These confounding conditions included, cardiac clinical symptoms or disease with left ventricular ejection fraction<50%, and hypertension that could not be well controlled with antihypertensive drugs.;
* All patients were assessed by the sarcoma board including a thoracic surgeon with at least 10 years surgical experience. Patients with lung metastases only were carefully assessed for eligibility for metastasectomy, of whom those who were suitable for surgery were excluded from this study;
* weight loss of 20% or more before illness;
* brain or leptomeningeal metastasis;
* surgical procedure or radiotherapy within 4 weeks of enrollment;
* activegastroduodenal ulcer, previous condition associated with risk of bleeding or requiring anticoagulation;
* proteinuria or hematuria, denutrition with albuminemia <25 g/L;
* women who were pregnant or breast feeding, other malignancy;
* positive HBV/HCV/HIV serology, and known allergy to the experimental agents.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 2 years
  from the start of target treatment until disease progression or death, whichever came first.

SECONDARY OUTCOMES:
Overall survival | 3 years
  from the date of treatment initiation to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Guo, M.D., Principal Investigator — Musculoskeletal Tumor Center of Peking University People's Hospital
Locations (2):
- China (2):
  - Peking University Shougang Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Undecided